CLINICAL TRIAL: NCT05781061
Title: Medication Abortion With Autonomous Self-Assessment Project at Independent Abortion Clinics: A Demonstration Project
Brief Title: MA-ASAP at Independent Abortion Clinics: A Demonstration Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: All Families Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1059
Record Dates: First submitted 2023-03-01; First posted 2023-03-23 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2023-03

CONDITIONS: Abortion Early
MeSH Terms: interventions — Mass Screening; Eligibility Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asynchronous Screening (Experimental): Participants will be screened for medication abortion eligibility using written or online materials and questionnaires, without a synchronous conversation between the prescribing clinician and the patient.
  Interventions: Other: Screening for Eligibility

INTERVENTIONS:
Other: Screening for Eligibility — Asynchronous Screening for MA Eligibility

SUMMARY:
In this study, the investigators propose to conduct a parallel study to MA-ASAP (ClinicalTrials.gov Identifier: NCT05278780) at an independent clinic.

DETAILED DESCRIPTION:
In this study, the investigators propose to conduct a parallel study to the MA-ASAP pilot study (ClinicalTrials.gov Identifier: NCT05278780) at one or more independent abortion clinics. This new study will be similar in structure to pilot study, except that all completed screening questionnaires will be sent to the study site rather than only those deemed eligible according a computer algorithm. The investigators expect that this change will better serve the needs of both clinics and patients, and it will also allow us to assess whether the algorithm is overly restrictive, i.e., whether it is excluding patients who are in fact eligible for MA. The primary goal of the study is to collect data on feasibility of the approach and safety. Secondarily, the investigators aim to assess the ability of a defined set of responses to the screening questionnaire to predict the clinician's decision about whether a clinical consultation is needed.

ELIGIBILITY:
Inclusion Criteria:

* Can speak and read English
* Has an address in a state where the study clinicians are licensed to practice medicine and where the service is legal
* Is old enough to consent to abortion and study participation without parental consent in the study state
* Has reviewed the study website
* Has had a positive pregnancy test
* Has signed the study informed consent form (ICF), which will be included within the questionnaire
* Is pregnant with a gestational age of ≤77 days from last menstrual period
* Desires MA
* Has no symptoms of or risk factors for ectopic pregnancy
* Has no medical contraindications to MA, specifically:

Hemorrhagic disorder or concurrent anticoagulant therapy Chronic adrenal failure Concurrent long-term systemic corticosteroid therapy Inherited porphyria Allergy to mifepristone or misoprostol, or other prostaglandin

* Is not asked by the site to have a synchronous consultation with clinician OR facility-based tests such as ultrasound, laboratory tests, examination, etc.
* Is comfortable obtaining the abortion pills without a pre-treatment ultrasound and without speaking by phone or video with the abortion provider.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of participant questions | 6 months
  The proportion of participants who have questions after completing the questionnaire and the types of questions that are asked.
Proportion of participants that are followed through the study | 6 months
  The numbers and proportions of people who complete the questionnaire once initiated, are reached by study staff after submitting a completed questionnaire, and are ultimately followed through the study.
Incidence of reported problems by site staff | 6 months
  Problems with the study process as reported by site staff
Study site satisfaction (self-reported) | 6 months
  Interest on the part of study sites to continue to utilize this approach to MA provision after the study ends.
Incidence of Treatment-Emergent Adverse Events | 6 months
  Proportion of treated participants with SAE related to the study

SECONDARY OUTCOMES:
Efficacy of computer algorithm to determine MA eligibility | 6 months
  We will estimate the predictive value of this algorithm for selecting participants who were deemed eligible for MA or ultimately did receive treatment without a synchronous consultation or facility-based tests

CONTACTS AND LOCATIONS:
Locations (1):
- All Families Healthcare, Whitefish, Montana, United States

IPD SHARING:
Plan to Share IPD: No